CLINICAL TRIAL: NCT00138528
Title: Other Effects of Fluvastatin Are Investigated in Patients With Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CXUO320BDE30
Record Dates: First submitted 2005-08-25; First posted 2005-08-30 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome, fluvastatin
MeSH Terms: conditions — Metabolic Syndrome | interventions — Fluvastatin

INTERVENTIONS:
Drug: Fluvastatin

SUMMARY:
Other effects of fluvastatin are investigated in German patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male and female patients, aged between 18 and 75 years
* Metabolic syndrome according to National Cholesterol Education Program Adult Treatment Panel III (NCEP ATPIII)

Exclusion Criteria:

* History of heart failure
* HIV positive
* Stroke

Other protocol defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2004-10; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in circulating marker of inflammation (C-reactive protein) after 5 weeks

SECONDARY OUTCOMES:
Change from baseline in low density lipoprotein cholesterol after 5 weeks
Change from baseline in non high density lipoprotein cholesterol after 5 weeks
Change from baseline in total cholesterol after 5 weeks
Change from baseline in high density lipoprotein cholesterol after 5 weeks
Change from baseline in oxidized low density lipoprotein cholesterol after 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Nuremberg, Germany

REFERENCES:
- [Result] Westphal S, Abletshauser C, Luley C. Fluvastatin treatment and withdrawal: effects on endothelial function. Angiology. 2008 Oct-Nov;59(5):613-8. doi: 10.1177/0003319708316005. Epub 2008 Apr 14. PMID 18413332